CLINICAL TRIAL: NCT01276119
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-center, Single-dose, Dose-escalating Study to Evaluate the Safety and Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of CDP6038 in Healthy Male Subjects
Brief Title: The First Clinical Study to Test Safety, Blood Levels and Other Effects of CDP6038 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: RA0001
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Pharmacokinetics
Keywords: CDP6038; single-dose; pharmacokinetics; healthy subjects
MeSH Terms: interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (14):
- Cohort A, CDP6038 0.001 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort B, CDP6038 0.01 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort C, CDP6038 0.03 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort D, CDP6038 0.1 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort E, CDP6038 0.3 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort G, CDP6038 1.0 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort I, CDP6038 3.0 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort K, CDP6038 10.0 mg/kg, iv (Experimental)
  Interventions: Biological: CDP6038
- Cohort A, Placebo, iv (Placebo Comparator)
  Interventions: Other: Placebo
- Cohort B, C, D, E, G, I, K, Placebo, iv (Placebo Comparator)
  Interventions: Other: Placebo
- Cohort F, CDP6038 0.3 mg/kg, sc (Experimental)
  Interventions: Biological: CDP6038
- Cohort H, CDP6038 1.0 mg/kg, sc (Experimental)
  Interventions: Biological: CDP6038
- Cohort J, CDP6038 3.0 mg/kg, sc (Experimental)
  Interventions: Biological: CDP6038
- Cohort F, H, J, Placebo, sc (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CDP6038 — 100 mg/mL solution for injection Single infusion over 60 minutes
  Arms: Cohort A, CDP6038 0.001 mg/kg, iv
Biological: CDP6038 — 100 mg/mL solution for injection Single infusion over 120 minutes
  Arms: Cohort B, CDP6038 0.01 mg/kg, iv; Cohort C, CDP6038 0.03 mg/kg, iv; Cohort D, CDP6038 0.1 mg/kg, iv; Cohort E, CDP6038 0.3 mg/kg, iv; Cohort G, CDP6038 1.0 mg/kg, iv; Cohort I, CDP6038 3.0 mg/kg, iv; Cohort K, CDP6038 10.0 mg/kg, iv
Biological: CDP6038 — 100 mg/mL solution for injection Single sc injection
  Arms: Cohort F, CDP6038 0.3 mg/kg, sc; Cohort H, CDP6038 1.0 mg/kg, sc; Cohort J, CDP6038 3.0 mg/kg, sc
Other: Placebo — 0.9% sodium chloride for injection Single infusion over 60 minutes
  Arms: Cohort A, Placebo, iv
Other: Placebo — 0.9% sodium chloride for injection Single infusion over 120 minutes
  Arms: Cohort B, C, D, E, G, I, K, Placebo, iv
Other: Placebo — 0.9% sodium chloride for injection Single sc injection
  Arms: Cohort F, H, J, Placebo, sc

SUMMARY:
To evaluate the safety, tolerability, blood levels and effects of CDP6038 administered by intravenous infusion (iv) and subcutaneous (sc) injection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 19.0 and 28.0 kg/m² and body weight between ≥ 50 kg and ≤ 120 kg

Exclusion Criteria:

* Previous trial participation or blood donation/loss within 3 months
* Subject is not healthy (eg significant medical history, taking drug treatments, any psychological or emotional problems, or drug or alcohol abuse (current or historical)
* Plans for or actual vaccination within 3 months
* Previous drug treatments
* Tobacco use or heavy caffeine consumption
* Systolic blood pressure <90 or >145mmHg, diastolic blood pressure <40 or >90mmHg or heart rate <45 or >90 beats per minute

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The maximum drug concentration (Cmax) of CDP6038 in plasma given by intravenous (iv) infusion and subcutaneous (sc) injection in healthy male subjects. | Baseline to 14 weeks
The area under the plasma concentration/time curve from hour 0 to the time with the last quantifiable level of CDP6038 given by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks
The area under the plasma concentration/time curve extrapolated to infinity, of CDP6038 given by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks
The half life of CDP6038 in plasma given by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks
The apparent volume of distribution of CDP6038 given by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks
Total body clearance of CDP6038 in plasma given by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks
PK/PD relationship between systemic CDP6038 exposure and suppression of selected acute phase markers (such as C-reactive protein) following CDP6038 administration by iv infusion and sc injection in healthy male subjects. | Baseline to 14 weeks

SECONDARY OUTCOMES:
Anti-CDP6038 antibodies in plasma following iv infusion and sc injection of CDP6038 in healthy male subjects. | Baseline to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Berlin, Germany